CLINICAL TRIAL: NCT04985682
Title: Phase 4, Multicenter, Prospective, Interventional, Post-Marketing Study in Hemophilia A Patients in India Receiving ADVATE as On-Demand or Prophylaxis Under Standard Clinical Practice
Brief Title: A Study of ADVATE in People With Hemophilia A in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-761-4009; 2022-004149-11 (EudraCT Number)
Record Dates: First submitted 2021-07-29; First posted 2021-08-02 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-08

CONDITIONS: Hemophilia A
Keywords: Drug Therapy
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemophilia A Group (Experimental): Participants with hemophilia A were treated with ADVATE according to a regimen determined by the treating physician at the study site and in accordance with the national product label under standard clinical practice for 6.7 months.
  Interventions: Biological: ADVATE

INTERVENTIONS:
Biological: ADVATE — Antihemophilic factor (AHF) activity expressed in international units (IU) per vial.

SUMMARY:
The main aim of this study is to learn more about side effects of Advate when given as standard treatment to people with hemophilia A who have already been treated.

The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study. Participants will need to visit the study doctor 5 times in total during the study. During these visits, study data will be collected by the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* The participant or legally authorized representative (in case of study participants less than (<) 18 years of age) gave written informed consent to participate in the study.
* Participant of any age with hemophilia A.
* Participant defined as a previously treated patient (PTP):

  * Participant aged greater than or equal to (>=) 6 years that has been previously treated with plasma-derived and/or recombinant FVIII concentrate(s) for a minimum of 150 exposure doses (EDs).
  * Participant aged less than <6 years that has been previously treated with plasma-derived or recombinant FVIII concentrate(s) for a minimum of 50 EDs.
* Participant as negative history of FVIII inhibitors and negative inhibitor at screening defined as less than 0.6 Bethesda units (BU) per milliliter (Nijmegen-modified Bethesda assay).
* Participant is human immunodeficiency virus negative (HIV-); or human immunodeficiency virus positive (HIV+) with stable disease and cluster of differentiation 4 (CD4+) count >=200 cells per cubic millimeter (mm^3), as confirmed by central laboratory at screening.
* Participant is hepatitis C virus negative (HCV-) by antibody or polymerase chain reaction (PCR) testing (if positive, anti-body titer will be confirmed by PCR), as confirmed by central laboratory at screening; or hepatitis C virus positive (HCV+) with chronic stable hepatitis.
* Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Participant has known hypersensitivity to mouse or hamster proteins or to any of the excipients of FVIII (factor VIII) concentrates.
* Participant has been diagnosed with bleeding disorder(s) other than congenital hemophilia A, such as acquired hemophilia A, von Willebrand´s disease (VWD) or thrombocytopenia (platelet count <100,000 per milliliter).
* Participant has received treatment for hemophilia A with non-FVIII products or concentrates (example, emicizumab [Hemlibra®]) in the 6 months prior to screening.
* Participant has severe chronic hepatic dysfunction (example, >=5 times upper limit of normal alanine aminotransferase [ALT], aspartate aminotransferase [AST] or international normalized ratio [INR] >1.5 as confirmed by central laboratory at screening).
* Participant has planned or is likely to have, surgery during the study period.
* Participant has a clinically significant medical, psychiatric, or cognitive illness, or recreational drug or alcohol use that, in the opinion of the investigator, would affect participant's safety or compliance.
* Participant currently receiving or is scheduled to receive during the course of the study, an immunomodulating drug (example, corticosteroid agents at a dose equivalent to hydrocortisone >10 milligram per day, or α-interferon) other than antiretroviral chemotherapy.
* Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
* Participant is a family member or employee of the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (5):
- India (5):
  - Amrita Institute of Medical Science & Research Centre, Ernākulam, Kerala
  - St. John's Medical College, Bengaluru
  - K J Somaiya Hospital & Research Centre, Mumbai
  - All India Institute of Medical Sciences (AIIMS), New Delhi
  - Unique Children's Hospital Pvt. Ltd., Pune

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61044886beb21d002a92608f

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in India from 14 January 2022 to 10 February 2023.
Pre-assignment Details: Participants previously treated for hemophilia A who met eligibility criteria were enrolled to receive ADVATE according to a dosing regimen determined by the treating physician and in accordance with the national product label.
Period: Overall Study
Arm/Group | Hemophilia A Group
Started | 50
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Effectiveness Full Analysis Set (EFAS) comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 50
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 50
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 48.5 (20.95)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 152.0 (22.68)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI = Weight (kg)/Height (m)^2
  kilograms per meter square (kg/m^2) | 19.9 (5.42)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAE) at Least Possibly Related to ADVATE
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this investigational product or medicinal product. An SAE was defined as any untoward medical occurrence that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of present hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or was a medically important event. Number of participants with SAEs (including FVIII inhibitor formation) that were at least possibly related to ADVATE were reported.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: Safety Analysis Set (SAS) included all participants who received ADVATE at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
Participants | 0

2. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) at Least Possibly Related to ADVATE
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this investigational product or medicinal product. Number of participants with non-serious AEs that were at least possibly related to ADVATE were reported.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: SAS included all participants who received ADVATE at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
Participants | 0

3. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included hematology, clinical chemistry, viral serology, factor VIII (FVIII) antigen, FVIII activity, incremental recovery, and FVIII inhibitor. Clinical significance was judged as per Investigator's assessment.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: SAS included all participants who received ADVATE at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
Participants | 0

4. Secondary Outcome: Total Annualized Bleeding Rate (ABR) With Prophylactic Treatment of ADVATE
Description: ABR was defined as number of bleeding episodes during the study period divided by total number of study period days multiplied by 365.25. The mean ABR and standard error was estimated using a generalized linear model (GLM). The total ABR is reported in this outcome measure.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Error); unit: bleeds per year
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
bleeds per year | 2.65 (0.195)

5. Secondary Outcome: ABR With Prophylactic Treatment of ADVATE Categorized Based on Location of Bleed
Description: ABR was defined as number of bleeding episodes during the study period divided by total number of study period days multiplied by 365.25. The mean ABR and standard error were estimated using a GLM. The ABR by bleed sites (example, joint, soft tissue, muscle, other [mouth, gums or nose] are reported in this outcome measure.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Error); unit: bleeds per year
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
bleeds per year
  Bleed Location: Joint | 2.33 (0.203)
  Bleed Location: Soft Tissue | 0.04 (1.000)
  Bleed Location: Muscle | 0.16 (0.628)
  Bleed Location: Other (Mouth, Gums or Nose) | 0.12 (0.813)

6. Secondary Outcome: ABR With Prophylactic Treatment of ADVATE Categorized Based on Type of Bleed
Description: ABR was defined as number of bleeding episodes during the study period divided by total number of study period days multiplied by 365.25. The mean ABR and standard error were estimated using a GLM. The ABR by bleed cause (example, spontaneous, injury, and unknown) are reported in this outcome measure.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Error); unit: bleeds per year
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
bleeds per year
  Bleed Type: Spontaneous | 1.86 (0.211)
  Bleed Type: Injury | 0.20 (0.692)
  Bleed Type: Unknown | 0.59 (0.541)

7. Secondary Outcome: Total Number of ADVATE Infusions Required During Prophylactic Treatment
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Deviation); unit: infusions
Groups:
- Haemophilia A Group: Participants with hemophilia A were treated with ADVATE according to a regimen determined by the treating physician at the study site and in accordance with the national product label under standard clinical practice for 6.7 months.
Arm/Group | Haemophilia A Group
Number analyzed (Participants) | 50
infusions | 65.8 (22.92)

8. Secondary Outcome: Average Number of ADVATE Infusions Required Per Week During Prophylactic Treatment
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Deviation); unit: infusions per week
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
infusions per week | 2.5 (0.87)

9. Secondary Outcome: Average Number of ADVATE Infusions Required Per Month During Prophylactic Treatment of Bleeding Episode
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Deviation); unit: infusions per month
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
infusions per month | 11.0 (3.76)

10. Secondary Outcome: Total Body Mass Adjusted Consumption of ADVATE During Prophylactic Treatment
Description: Body mass adjusted consumption international units per kilograms (IU/kg) was derived as the total units infused (IU) divided by the last available body weight (kg) prior to the infusion.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
IU/kg | 1739.7 (621.18)

11. Secondary Outcome: Average Body Mass Adjusted Consumption of ADVATE Per Week During Prophylactic Treatment
Description: Body mass adjusted consumption (IU/kg) was derived as the total units infused (IU) divided by the last available body weight (kg) prior to the infusion.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Deviation); unit: IU/kg per week
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
IU/kg per week | 67.1 (24.12)

12. Secondary Outcome: Average Body Mass Adjusted Consumption of ADVATE Per Month During Prophylactic Treatment
Description: as for outcome 11
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met.
Measure: Mean (Standard Deviation); unit: IU/kg per month
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 50
IU/kg per month | 291.7 (104.80)

13. Secondary Outcome: Overall Hemostatic Efficacy Rating of ADVATE for Treatment of Bleeding Episodes
Description: Overall hemostatic efficacy for treatment of bleeding episodes was rated on 4-point Likert scale as: excellent=full relief of pain and cessation of objective signs of bleeding after a single infusion, no additional infusion is required for the control of bleeding and administration of further infusion to maintain hemostasis would not affect the scoring; good=definite pain relief and/or improvement in signs of bleeding after a single infusion, possibly requires more than 2 infusions for complete resolution and administration of further infusion to maintain hemostasis would not affect the scoring; moderate=probable and/or slight relief of pain and slight improvement in signs of bleeding after a single infusion, required multiple infusions for complete resolution; none=no improvement of signs or symptoms or conditions worsen.
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: EFAS comprised of all participants for whom all inclusion and none of the exclusion criteria were met. Overall number of participants analyzed are the number of participants with bleeds who required ADVATE infusion for management of the bleeding episode.
Measure: Number; unit: bleeding episodes
Units Other Than Participants: Treated Bleeds
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 24
Number analyzed (Treated Bleeds) | 51
bleeding episodes
  Excellent | 21
  Good | 26
  Moderate | 4
  None | 0

14. Secondary Outcome: Number of ADVATE Infusions Required to Achieve Resolution of Bleeding Episodes
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 24
infusions | 1.2 (0.46)

15. Secondary Outcome: Total Body Mass Adjusted Consumption of ADVATE Per Bleeding Episode
Description: as for outcome 11
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Hemophilia A Group
Number analyzed (Participants) | 24
IU/kg | 34.8 (19.79)

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) up to end of study (up to 12.9 months)
Description: SAS included all participants who received ADVATE at any time during the study.
Arm/Group | Hemophilia A Group
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 6/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemophilia A Group (N=50)
Pyrexia (General disorders) | 2 (2)
Varicella (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (3)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT04985682/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT04985682/SAP_001.pdf